CLINICAL TRIAL: NCT01962467
Title: A Relative Bioavailability Study to Compare the Pharmacokinetics of a Fixed Dose Combination of Fluticasone Furoate and Levocabastine With Levocabastine and Fluticasone Furoate Alone
Brief Title: A Relative Bioavailability Study of Fluticasone Furoate and Levocabastine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200284
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Rhinitis, Allergic, Perennial and Seasonal
Keywords: Allergic rhinitis; healthy volunteers; fluticasone furoate; levocabastine; fixed dose combination; pharmacokinetics
MeSH Terms: conditions — Rhinitis; Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Each subject will receive 7 once daily doses of one of the 3 treatments (FF/LEV FDC or FF or LEV) administered as two 50 µL sprays per nostril in the morning, during each of the 3 treatment periods, as per one of the 6 possible randomization sequences. Each treatment period will be separated by a minimum washout period of 14 days
  Interventions: Drug: FF/LEV FDC; Drug: FF; Drug: LEV

INTERVENTIONS:
Drug: FF/LEV FDC — Intranasal aqueous microsuspension containing 25.0 microgram (µg) of FF and 50 µg of LEV as a fixed dose combination. It will be administered as two 50 µL sprays per nostril in the morning in a fasted state
Drug: FF — Intranasal aqueous microsuspension containing 27.5µg of FF. It will be administered as two 50 µL sprays per nostril in the morning in a fasted state
Drug: LEV — Intranasal aqueous microsuspension containing 50 µg of LEV. It will be administered as two 50 µL sprays per nostril in the morning in a fasted state

SUMMARY:
This is an open label, randomized, 3-way cross-over, and repeat administration study in healthy male and female subjects. The purpose of the study is to determine the relative bioavailability of Fluticasone Furoate (FF) and Levocabastine (LEV), when each is administered alone and as FF/LEV Fixed Dose Combination (FDC).This study consists of Part A (in which 30 subjects including 12 Korean subjects will be enrolled) and Part B (in which 18 subjects will be enrolled). Each part will consist of three treatment periods separated by a minimum washout period of 14 days. In each treatment period, subjects will receive seven daily doses of one of the 3 treatments: FF, LEV or FF/LEV FDC, via an intranasal spray according to one of the 6 possible randomization sequences. The study will use an adaptive design with an interim review following Part A to confirm whether Part B is required.

ELIGIBILITY:
Inclusion Criteria:

* Male/Females aged between 18, 20 for Korean subjects, and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Caucasian, defined as having four grandparents who were descendents of European Caucasians, or Korean origin defined as being born in mainland Korea, having four ethnic Korean grandparents, holding a Korean passport or identity papers and being able to speak Korean. Korean subjects should also have lived outside their respective countries for less than 10 years.
* Body weight >=50 kilogram (kg), >=45 kg for Korean subjects, and body mass index (BMI) within the range 18 - 30 Kilogram per meter square (kg/m^2) (inclusive).
* A female subject is eligible to participate if she is of: non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy [for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records]; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli-international units per milliliter (MIU/mL) and estradiol <40 picogram/milliliter (pg/mL) (<147 picomole/liter) is confirmatory]; child-bearing potential with negative pregnancy test as determined by urine Human Chorionic Gonadotropin (hCG) test at screening or prior to dosing AND agrees to use one of the contraception methods as described for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 8 days post-last dose.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin <=1.5 x Upper Limit of Normal (ULN) [isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%].
* Based on single or averaged corrected QT interval (QTc) values of triplicate electrocardiograms (ECGs) obtained over a brief recording period: QT interval corrected for heart rate using Fridericia'sformulas (QTcF) <450 milliseconds (msec).

Exclusion Criteria:

* Criteria Based Upon Medical Histories:
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of regular alcohol consumption within 6 months of the study defined as: For Australian (AUST) sites: An average weekly intake of >21 units for males or > 14 units for females. In Australia one unit (=standard drink) is equivalent to 10 grams (g) of alcohol: 270 mL of full strength beer (4.8%), 375 mL of mid strength beer (3.5%), 470 mL of light beer (2.7%), 250 mL pre-mix full strength spirit (5%), 100 mL of wine (13.5%) and 30 mL of spirit (40%).
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation.
* Nasal abnormalities likely to affect the outcome of the study, i.e., nasal septal perforation, nasal polyps, other nasal malformations.
* History of frequent nosebleeds.
* Subjects should be non-smokers, which for this study is defined as having smoked < 10 pack years in their lifetime, and have not smoked in the 6 months prior to the screening visit.

Criteria Based Upon Diagnostic Assessments

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* A positive pre-study drug/alcohol screen.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Urine cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Other Criteria:
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Lactating females.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Any history of nasal surgery which may affect the outcome of the study (i.e., turbinectomy, major nasal reconstruction, septal perforation repair).
* Any history in the past 5 years of either perennial or seasonal allergic rhinitis, or any subject expected to have symptoms of allergic rhinitis during the study.
* Subjects with recent upper respiratory tract infections (URTIs) will be allowed in the study only if their nasal symptoms associated with the URTI have been completely resolved for more than 3 weeks prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-10-11 (Actual); Primary Completion 2014-02-27 (Actual); Study Completion 2014-02-27 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of FF and LEV | Day 7 (Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose) and Day 8 (24 hours post-dose) of each treatment period
  Concentrations of FF and LEV will be determined in plasma samples
Pharmacokinetic (PK) parameters for both FF and LEV | Day 7 (Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose) and Day 8 (24 hours post-dose) of each treatment period
  From the plasma concentration-time data, area under the plasma concentration-time curve (AUC) and maximum plasma concentration (Cmax) of FF and LEV were determined

SECONDARY OUTCOMES:
PK parameters for both FF and LEV alone and in combination | Day 7 (Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose) and Day 8 (24 hours post-dose) of each treatment period
  From the plasma concentration-time data, AUC, Cmax and time to maximum observed plasma drug concentration (tmax) of FF and LEV alone and in combination were determined for healthy Korean male and female subjects
tmax | Day 7 (Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 6, 8, and 12 hours post-dose) and Day 8 (24 hours post-dose) of each treatment period
  Tmax of FF and LEV alone and in combination were determined for healthy male and female subjects

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 200284 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/200284?search=study&search_terms=200284#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 200284 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200284 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200284 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200284 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200284 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200284 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200284 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register